CLINICAL TRIAL: NCT03981302
Title: Family Nursing Conversations With Patients With Chronic Non-cancer Pain and Their Selected Family Members. Protocol for the FANCOC-PAIN Quasi-experimental Trial
Brief Title: Family Nursing Conversations Patients With Chronic Non-Cancer Pain
Acronym: FANCOC-PAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bente Appel Esbensen (Other)
Collaborators: Rigshospitalet, Denmark (Other); University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Bente Appel Esbensen, Research Manager and Associate Professor, Glostrup University Hospital, Copenhagen
Organization: Glostrup University Hospital, Copenhagen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Family nursing chronic pain
Record Dates: First submitted 2019-06-04; First posted 2019-06-10 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Chronic Nonmalignant Pain
Keywords: Chronic Nonmalignant Pain; Family Nursing; Multidisciplinary Pain Center; Quasi-Experimental Study

STUDY DESIGN:
Intervention Model Description: The study has a quasi-experimental design and will conduct baseline and post-test in two comparable groups of patients and their selected family members: An intervention group and a historical control group. The data from the historical control group will be collected initially in the study to prevent pollution of the data when the intervention nurses are educated in Family nursing.
  The study is a part of a superior explanatory sequential mixed methods design consisting of a total of three substudies. The two other substudies have qualitative designs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family nursing conversations (Experimental): The intervention will consist of structured family nursing conversations between a nurse, the patient and their selected family members. The patients will receive the intervention and usual treatment.
  Interventions: Other: Family nursing conversations
- Usual treatment (No Intervention): The patients will receive usual treatment.

INTERVENTIONS:
Other: Family nursing conversations — The intervention is based on the concept "family systems nursing" developed by Wright & Maureen. Family nursing aims to change restricting beliefs and alleviate illness suffering. The Illness Beliefs model and Calgarymodels are essential components. The illness beliefs model illuminates the family's different beliefs about their problems. The Calgary models consist of the Calgary family assessment model and the Calgary intervention model and aim to support change and help the family to find new ways to handle the illness. The use of the components cannot be standardised but must be tailored to match the needs of the specific family. The family nursing conversations in this intervention will last 1,5 hour. Every family will be offered three family nursing conversations with roughly three weeks interval. If the family after three conversations express a need for follow-up, they will be offered the fourth conversation.
  Arms: Family nursing conversations

SUMMARY:
This study assumes that family nursing will enhance the management of chronic nonmalignant pain (CNP) for the patients and their family members. CNP accounts for a major healthcare problem with a thorough impact on several levels. Living with CNP is a condition of life, that calls for acceptance, but due to the invisible nature of CNP, the patients often experience a lack of understanding and doubt about the condition´s reality making acceptance challenging. Research indicates that the involvement of relatives has a positive effect on the management of CNP. An existential need for individualised adapted involvement is expressed by patients and relatives. Family nursing has the potential to comply with the expressed need but is not investigated on patients with CNP.

The objective of the study is to explore if an intervention with systematic family nursing conversations with patients with chronic nonmalignant pain and their selected family members is effective on primary self-efficacy and secondary family function, quality of life and anxiety/depression. The intervention is based on the concept of "family systems nursing" developed by Wright and Leahey. Besides usual treatment, the intervention consists of 3-4 structured conversations each 1,5 hour between the nurse, the patient and their selected family members. Previous to the intervention, the involved nurses will go through a family nursing course of three days duration. During the intervention, regular reflection sessions will be conducted.

The study design is quasi-experimental with a baseline- and a post-test in two comparable groups of patients and their selected family members: An intervention group and a control group. The design is chosen to prevent contamination of the control group data if the nurses change behaviour regarding families after participating in the course. Collection of data from the control group will be completed before the course. In the intervention group, a follow-up assessment will be conducted four months after the post-test. Structured telephone interviews will obtain the selected self-reported outcomes from patients and their family members.

The study will follow the ethical guidelines of the Declaration of Helsinki (World-Medical-Association, 2008). The Data Protection Agency has approved the study with j-number VD-2019-152. According to The Danish National Committee on Health Research Ethics, there is no obligation to notify the study (record number: H-19016896).

DETAILED DESCRIPTION:
Introduction

This study assumes that family nursing for the patients with Chronic nonmalignant pain (CNP) and their family members by increased self-efficacy will enhance the management of the changed life condition and alleviate the related suffering of the family. The study has a quasi-experimental design and is the first sub-study of a superior mixed methods study consisting of a total of three sub-studies. The other substudies apply qualitative designs.

Background

CNP is usually understood as pain with a duration of at least three months with no relation to life-threatening causes. CNP accounts for a major healthcare problem with a thorough impact on several levels. Nineteen per cent of the adult European population has been found to suffer from moderate to severe CNP, which decreases physical and mental health, ability to work, wellbeing and quality of life. Additional mortality is increased. CNP has consequences for the patients´ social network as well and is associated with a poorer family function. The relatives get affected themselves with reduced physical and mental health. Living with CNP is a condition of life, that calls for acceptance. But CNP is an invisible illness, and despite the considerable impact, the patients often experience a lack of understanding and doubt about, whether the CNP is real. In the strive to achieve a legitim sick role and help to alleviate the suffering, patients with CNP continually seek out the health care system. The expenses at the socioeconomic level are compared to other chronic diseases comprehensive. Thus, gaining acceptance of CNP may be challenging.

Involvement of relatives for patients with CNP is sparsely described in the literature, but indicates, that involvement increases marital satisfaction and contribute to a better outcome for both patients and spouses. Managing CNP necessitates "being on the same page", and involvement of relatives is vital to obtain a common understanding. Within other disease areas, the involvement of relatives has resulted in reduced stress for spouses, closer family relations and increased family function. Thus, it may be assumed that the involvement of relatives has a positive effect on the management of CNP.

A multicenter study exploring experiences, needs and preferences of the patient, relatives and pain specialists regarding the involvement of relatives in chronic pain trajectories indicates that patients and relatives have an existential need for individualised adapted involvement. Family nursing based on the concept of "family systems nursing" developed by Lauren Wright and Maureen Leahey has the potential to comply with the expressed need. Wright and Leahey´s understanding of family nursing is inspired by the postmodernism and biology of cognition and based on theories of systems, communication, cybernetic and change. The nurse must simultaneously concentrate on both patient and family and focus on interaction, reciprocity and connection between different systems, consisting of the patient, the family and the larger system they are a part of. Family nursing aims to change restricting beliefs and alleviate illness suffering. The essential components of the family systems nursing concept comprise the clinical practice models: The Illness Beliefs model and the Calgarymodels. The illness beliefs model illuminates the family's different beliefs about their problems. The Calgary models consist of the Calgary family assessment model and the Calgary intervention model and aim to support change and help the family to find new ways to handle the illness. In the family assessment, the nurse may use the concrete assessment tools: Genogram and ecomap to draw the internal and external structures of the family. The intervention model is focusing on strength and resilience in the family instead of deficits and dysfunction and describes the cognitive, affective and behavioural interventions the nurse may use to facilitate change. Family nursing and the clinical practice models are operationalised within a therapeutic relationship between the nurse, the patient and the family members, making the conversation fundamental to perform family nursing. Using questions during the conversations is essential to create new perspectives and alleviate suffering. Questions may provide information for both the nurse and the family, and an invitation to tell about illness experiences may on its own be a healing intervention. There is a distinction between two kinds of questions making a dichotomy. Assessment/linear questions are investigating and intend to provide information for the nurse. Interventional/circular questions invite to reflection, initiate change and encourage the family members to understand their problems in new ways and find new solutions.

The rationale of the study

Summarised CNP is a condition with radical consequences on several levels. Due to the chronicity of the condition, management is necessary, but the impact and invisibility of CNP impede this discipline. It is assumed that the involvement of relatives will strengthen patient's and family members self-efficacy and benefit the process of acceptance. Family nursing based on the family systems nursing concept has the potential to comply with the need for individualised adapted involvement expressed by patients and relatives but has not been investigated on patients with CNP. Family nursing interventions in other illness areas have shown positive. An integrative review describing the reactions from diseased families, who participated in family nursing interventions finds that the family response corresponds to the intention of family nursing. However, there is a need for further illness specific and quantitative research since existing knowledge primary is based on qualitative studies.

Aim

The objective of this study is to investigate, whether an intervention with systematic conversations with patients with chronic nonmalignant pain and their selected family members in a context of family nursing is effective on primary self-efficacy and secondary family function, quality of life and anxiety/depression.

Setting

The study will be conducted at the Multidisciplinary Pain Centre, Department of Neuroanaesthesiology, The Neuroscience Centre, Rigshospitalet, University of Copenhagen.

The intervention

The intervention with family nursing is based on the previously described concept of "family systems nursing". The intervention will consist of structured conversations named "family nursing conversations" between the nurse, the patient and up to three selected family members on 15 years or older. In the framework of family systems nursing the family is widely understood as a group of individuals who are bound by strong emotional ties, a sense of belonging, and a passion for being involved in one another's life. Thus, the notion of family members goes beyond relationships connected by law or genetic. Family nursing will, during the conversations, be operationalised by the selected components from the concept. The specific use of the components cannot be standardised since family nursing must be tailored to match the needs of the specific family. Each conversation takes 1,5 hour. Every family are offered three or four family nursing conversations as needed with roughly three weeks interval. All patients also receive the usual treatment from the Multidisciplinary Pain Centre. Previous to the intervention, the involved nurses will go through a three days family nursing course, and will during the intervention participate in regular reflection sessions.

Study design

The study design is quasi-experimental with a baseline- and a post-test in two comparable groups of patients and their selected family members: An intervention group and a control group. In the intervention group, a follow-up assessment will be conducted four months after the post-test. The design is chosen because the number of nurses in the chosen clinical setting is limited. All the nurses must participate in the family nursing course and will subsequently likely change their behaviour regarding the involvement of family members. The control group will be recruited at the beginning of the study to prevent contamination of data when the nurses' after the course have developed competencies to care for the whole family.

Outcomes and missing data

Structured telephone interviews will obtain the selected self-reported outcomes from patients and their family members. By this, the amount of missing data is expected to be minimal. All participants consisting of the patients and their selected family members are assessed by the same outcome measures. The primary outcome is General self-efficacy scale (GSE), and secondary outcomes are Iceland-Expressive Family Functioning Questionnaire (ICE-EFFQ), quality of life (SF12) and the Hospital Anxiety and Depression Scale (HADS). The study comprises a self-designed questionnaire for the patients and their family members with the chosen outcomes, socio-demographic data and health information.

Sample size

The sample size is based on the primary outcome GSE and the results from Scholz et al. 20002 regarding psychometric findings from 25 countries, including Denmark. Based on the average GSE on 29,716, with a significance level on 95% (α = 5), a power on 80 % (β = 20), a desired MIREDIF on 15% between the control group and the intervention group plus a calculated drop out on 25%, the sample size is calculated to 25 patient/family dyads in each group. Thus, a total of 50 patient/family dyads must be included. A patient/family dyad consists of one patient and a maximum of three selected family members. If the patient drops out, the entire dyad drops out. If a family member drops out, the dyad is retained in the project, when at least one family member continues. If all family members drop out, the dyad drops out as well.

Analysis

Data will be described from the selected questionnaires using conventional descriptive statistics, parametric statistics as regards normally distributed variables and non-parametric statistics as regard variables, that differs from the normal distribution. Logistic regression analyses are carried out to describe GSES-10, ICE-EFFQ, SF12, and HADS for patients and family members, who receive family nursing conversations and usual treatment. These are compared to patients and family members, who only receive usual treatment. Connections to socio-demographic data and health information will be described. The reporting of the study will attempt to meet the recommendations from The Joanna Briggs Institute Checklist for Quasi-Experimental Studies (non-randomized experimental studies).

Ethical

The study will follow the ethical guidelines of the Declaration of Helsinki. The study has been reported to the Data Protection Agency and is approved with j-number VD-2019-152. According to The Danish National Committee on Health Research Ethics, there is no obligation to notify the study (record number: H-19016896). The patients and their family members will receive written and oral information about the project according to the guidelines from the Danish National Committee on Health Research Ethics and rules about time to think it over will be followed. Written consent will be obtained, and verbal consent will be obtained before each telephone interview. Data will be anonymised throughout the analysis process and in all forms of reporting of the results. The aim is to include at the maximum three family members of each patient, but if the patient caused by this is forced to choose between the family members, the number of family members may be adjusted. Likewise, children younger than 15 years may be included, if it is considered proper and unethical to refrain from doing it.

ELIGIBILITY:
Inclusion Criteria:

* Patients who start a trajectory at the Multidisciplinary Paincentre at Rigshospitalet.
* Every patient selects a maximum of three family member at the age of 15 years or older, whom the patient from a comprehensive understanding perceive as a family

Exclusion Criteria:

* Patients or family members, who already receive family therapy with each other.
* Patients or family members, who are cognitively impaired.
* Patients or family members or dont speak or understand Danish.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
The general self-efficacy scale (GSE) | Assesed at week 9
  General self-efficacy refers to global confidence in one´s coping ability across a wide range of demanding or novel situations. GSE is tested in 25 countries, including Denmark, and GSE is suggested to be a universal construct. GSE consists of ten items with every four categories of answers varying from "not at all true" to "exactly true". Thus the score can range from 10 to 40. The higher the score, the higher the general self-efficacy. The average GSE is 29,716, but there is no cut-off score.

SECONDARY OUTCOMES:
Iceland-Expressive Family Functioning Questionnaire (ICE-EFFQ) | Assesed at week 9
  ICE-EFFQ is developed by the conceptual framework of Calgary Family Assessment Model for families, who experience acute or chronic illness. ICE-EFFQ measure family function within the last four weeks and consists of 17 items within four categories: Expressing emotions, collaboration and problem-solving, communication and behaviour. It uses a Likert scale with a scoring range from 1 (almost never) to 5 (all the time). The score can vary between 17 and 85. A high score indicates a good family function, but no exact cut-off score distinguishes between optimal or less optimal family function.
Quality of life, QoL (SF12) | Assesed at week 9
  SF-12 is the short form of a generic international quality of life instrument with 12 items, often used to asses health results and health-related quality of life. SF-12 measures self-reported health-related physical and mental quality of life. The SF12 provides data within the two main categories: Physical and mental health, each divided into four health domains. The total raw scores in each health domain are transformed into 0-100 scores, again transformed into T-scores. A higher score indicates a better health state.
The Hospital Anxiety and depression Scale (HADS) | Assesed at week 9
  HADS is developed to measure anxiety and depression in general medical outpatient clinics and takes into account that psychological and biological symptoms by medical diseases are hardly distinguishable. HADS consists of two subscales for respectively anxiety and depression with every seven items and measures self-reported symptoms the last seven days. The items are rated on a four-point scale and scored from 0-3 with total scores in each subscale ranging from 0-21. Scores between 0-7 represent no case, scores between 8-10 indicates mild cases, scores between 11-15 indicates moderate cases, and scores from 16 and above suggests severe cases.

CONTACTS AND LOCATIONS:
Overall Officials: Bente A Esbensen, Ass Prof, Principal Investigator — Rigshospitalet, Centre for rheumatology and spine diseases, copecare
Locations (1):
- Multidisciplinary Pain Centre, Department of Neuroanaesthesiology, The Neuroscience Centre, Rigshospitalet, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Full dataset to replicate the analysis will be available from the corresponding author on reasonable request until five years after completion of the study, according to Danish law.

REFERENCES:
- [Background] Reid KJ, Harker J, Bala MM, Truyers C, Kellen E, Bekkering GE, Kleijnen J. Epidemiology of chronic non-cancer pain in Europe: narrative review of prevalence, pain treatments and pain impact. Curr Med Res Opin. 2011 Feb;27(2):449-62. doi: 10.1185/03007995.2010.545813. Epub 2011 Jan 3. PMID 21194394
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. A classification of chronic pain for ICD-11. Pain. 2015 Jun;156(6):1003-1007. doi: 10.1097/j.pain.0000000000000160. No abstract available. PMID 25844555
- [Background] Bell JM. Family Systems Nursing: re-examined. J Fam Nurs. 2009 May;15(2):123-9. doi: 10.1177/1074840709335533. No abstract available. PMID 19423766
- [Background] Bell JM, Wright LM. The Illness Beliefs Model: advancing practice knowledge about illness beliefs, family healing, and family interventions. J Fam Nurs. 2015 May;21(2):179-85. doi: 10.1177/1074840715586889. No abstract available. PMID 25995203
- [Background] Ostlund U, Persson C. Examining Family Responses to Family Systems Nursing Interventions: An Integrative Review. J Fam Nurs. 2014 Aug;20(3):259-286. doi: 10.1177/1074840714542962. Epub 2014 Jul 15. PMID 25026964
- [Background] Chesla CA. Do family interventions improve health? J Fam Nurs. 2010 Nov;16(4):355-77. doi: 10.1177/1074840710383145. PMID 21051754
- [Background] Morales-Espinoza EM, Kostov B, Salami DC, Perez ZH, Rosalen AP, Molina JO, Gonzalez-de Paz L, Momblona JMS, Areu JB, Brito-Zeron P, Ramos-Casals M, Siso-Almirall A; CPSGPC Study Group. Complexity, comorbidity, and health care costs associated with chronic widespread pain in primary care. Pain. 2016 Apr;157(4):818-826. doi: 10.1097/j.pain.0000000000000440. PMID 26645546
- [Background] Glenton C. Chronic back pain sufferers--striving for the sick role. Soc Sci Med. 2003 Dec;57(11):2243-52. doi: 10.1016/s0277-9536(03)00130-8. PMID 14512253
- [Background] Swift CM, Reed K, Hocking C. A new perspective on family involvement in chronic pain management programmes. Musculoskeletal Care. 2014 Mar;12(1):47-55. doi: 10.1002/msc.1059. Epub 2013 Oct 7. PMID 24123548
- [Background] West C, Usher K, Foster K, Stewart L. Chronic pain and the family: the experience of the partners of people living with chronic pain. J Clin Nurs. 2012 Dec;21(23-24):3352-60. doi: 10.1111/j.1365-2702.2012.04215.x. Epub 2012 Jul 27. PMID 22834990